CLINICAL TRIAL: NCT06198868
Title: Minimal Residual Disease (MRD) Guided Prognosis Prediction and Adjuvant Treatment Based on Expression and Mutational Signatures of Circulating Tumor Cell (CTC) and Circulating Tumor DNA (ctDNA) in Non-small Cell Lung Cancer
Brief Title: MRD-guided Prognosis Prediction and Adjuvant Treatment Based on CTC and ctDNA in NSCLC
Status: Recruiting | Type: Observational
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Rong Yin, MD PhD, Professor, Jiangsu Cancer Institute & Hospital
Other Study IDs: 2023K-011
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Minimal Residual Disease; Prognosis monitoring; Adjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operable group: Early-stage patients with radical surgery or operable patients with neoadjuvant treatment
  Interventions: Procedure: Operable
- Inoperable group: Advanced-stage patients receive non-surgery therapies.

INTERVENTIONS:
Procedure: Operable — Enrolled patients capable of surgical treatment
  Groups: Operable group

SUMMARY:
This is a prospective cohort study, which aims to evaluate the effectiveness and superiority of a novel minimal residual disease-guided prognosis monitoring and adjuvant treatment in stage IIA-IIIC non-small cell lung cancer.

DETAILED DESCRIPTION:
This observational study is a single-center, prospective cohort study, which aims to detect minimal residual disease (MRD) using circulating tumor cells (CTC) and circulating tumor DNA (ctDNA). To evaluate the effectiveness and superiority of MRD detection, we enroll operable or inoperable IIA-IIIC stage NSCLC patients, and single-cell RNA sequencing and genomic sequencing would be performed for CTC and ctDNA, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed before implementing any enrollment-related procedures;
2. Age ≥18 years old;
3. Patients with histologically or cytologically confirmed stage IIA-IIIC NSCLC (International Association for the Study of Lung Cancer and American Joint Committee on Classification of Cancer, 8th Edition TNM staging)；
4. There is no special restriction on the source of genetic test report.
5. According to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1), there is at least one radiographically measurable lesion.
6. Have not received any previous systemic antitumor therapy for advanced diseases.
7. No serious abnormalities of hematopoietic function, heart, lung, liver, kidney function and immune system.
8. ECOG score: 0-1;
9. Expected survival time > 3 months.

Exclusion Criteria:

1. Received surgical treatment for lung tumors.
2. Received neoadjuvant chemotherapy or radiotherapy.
3. Received cellular therapy within the last 1 year.
4. Treated but uncontrolled diabetes, mellitus, asthma, autoimmune diseases and other chronic diseases.
5. Participated in other clinical trials (including research vaccines, drugs, medical devices, etc.) within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 patients with histologically or cytologically confirmed stage IIA-IIIC NSCLC would be enrolled from Jiangsu Cancer Institute & Hospital. In resectable group, we would enroll 20 early-stage cases and 20 operable patients for neoadjuvant treatment . In non-resectable group, 20 advanced-stage inoperable patients would be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Progression-free Survival (PFS) | From the first study dose date to the date of first documentation of disease progression or death (whichever occurred first), up to approximately 3 years
  Progression-free survival (PFS) is defined as the time from the start of treatment to the occurrence of tumor progression or death due to any cause based on RECIST 1.1 assessed by investigator review.

SECONDARY OUTCOMES:
To evaluate the Overall Survival (OS) | From the date of first dose of study drug until date of death from any cause (up to approximately 5 years )
  Overall Survival (OS) was measured from the date of first dose of study drug until date of death from any cause. Participants who were lost to follow-up and the participants who were alive at the date of data cutoff was censored at the date the participant was last known alive, whichever came earlier.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No